CLINICAL TRIAL: NCT01795794
Title: Evaluation of the Efficacy in Decreasing Iron Absorption in Patients With Congenital Dyserythropoietic Anemia Type I by Treatment With LOSEC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sor034612ctil
Record Dates: First submitted 2013-02-11; First posted 2013-02-21 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: CDA Type I
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LOSEC (Experimental): LOSEC will be given 20 mg X 1/day for 6 months and then for the next 6 months the same group will be the "control" group of herself.
  Interventions: Drug: omeprazole

INTERVENTIONS:
Drug: omeprazole
  Other Names: losec

SUMMARY:
Congenital Dyserythropoietic Anemia Type I (CDAI) is a recessive autosomal disease caused by ineffective erythropoiesis that causes Anemia & accumulation of iron due to increased absorption of iron in the intestine.

The iron is being accumulated in the body & causes damage of the liver, heart & endocrine glands.

The standard follow up of iron levels is done by ferritin blood test & although the test is not accurate it is the most available.

Medical treatment to removal of iron excess from the body is given in ferritin levels of 500-1000.

3 drugs are approved in the market:

* Deferoxamine, given subcutaneous during the night, 5-7 nights/week and therefore is less used today.
* Deferiprone-given 3 times a day, is a weaker chelator, although it seems like it is good to give it in combination with one of the 2 other drugs because it removes the iron from the heart's cells better.

A rare but severe adverse effect is Agranulocytosis. This drug is usually not given in childbirths.

-The 3rd drug which is mostly in use today is Deferasirox, given once daily, but has also adverse effects, among them- damage of liver & kidney function, damage to the digestive system, hearing and seeing.

Iron is being absorbed in acidic area, & thus drugs which decrease the acidity like hydrogen pump's inhibitors, can inhibit the absorption of iron, and indeed there are reports that these drugs decrease the absorption of iron and were used as treatment to hemochromatosis as well.

Those hydrogen pump's inhibitors have also adverse effects. The rarest but most severe is intestine infection by Clostridium.

In children, reports of adverse effects are minimal- mostly headaches & abdominal pains and nosocomial infections. In adults, there are reports of fractures, magnesium deficiency & vitamin B12 deficiency. All in all, the adverse effects are rare & uncommon.

DETAILED DESCRIPTION:
The aim of this study is to check whether treatment with drug which inhibits the hydrogen pump and therefore decreases acidity, will reduce the iron's absorption in patients with CDA TYPE I and whether it will be possible to use it for a period instead of giving drugs which have much more adverse effects, for removal of iron excess from the body.

Therefore, we would like to enroll 10-12 patients over 30 kg who can swallow tablets (age over 12) and whose ferritin levels are higher from the normal range, but still don't require medical treatment (ferritin levels between 400-700).

These patients will be given LOSEC 20 mg X 1/day for 6 months. That group will be her own control group in the 6 months later. Drug will be dispensed to the patients.

In the beginning of the study, after signing Informed Consent Form, blood tests will be taken for Complete Blood Count, iron levels, iron saturation, ferritin, complete chemistry panel, including calcium & magnesium.

Same tests will be taken after 3 and 6 months and also 3 and 6 months after end of treatment.

In every event of fever, headaches, abdominal pain or diarrhea, patients need to apply the doctor and report.

ELIGIBILITY:
Inclusion Criteria:

* patients with CDAI
* over 30 kg
* can swallow tablets
* ferritin levels higher than the normal range but still don't require treatment.

Exclusion Criteria:

* N.A

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
evaluate number of adverse effects per patient treated with LOSEC + levels of iron, ferritin,complete blood count and chemistry panel. | 1 year